CLINICAL TRIAL: NCT07365020
Title: A Feasibility Randomised Controlled Trial of Culturally Appropriate Physical Activity Promotion Strategies Among Older Chinese Adults in the UK
Brief Title: Feasibility RCT of Culturally Appropriate Physical Activity Strategies for Older Chinese Adults in the UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Yang Yang, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-19749-37005
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity; Ethnic Minority Group
Keywords: physical activity; ethnic minority group; intervention; randomised control trial; older Chinese adults; UK; Feasibility
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a culturally appropriate physical activity promotion strategies group or a control group receiving standard WHO physical activity information and are followed in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The culturally appropriate physical activity promotion strategies (Experimental): The culturally appropriate physical activity promotion strategies were developed based on 27 BCTs and will be delivered through three parts: a series of booklets, three workshops and a virtual social media support group
  Interventions: Behavioral: The culturally appropriate PA promotion strategies
- WHO physical activity guideline group (Active Comparator): The printed leaflet of recommendations from the WHO physical activity guideline for older adults
  Interventions: Behavioral: WHO leaflet group (control)

INTERVENTIONS:
Behavioral: The culturally appropriate PA promotion strategies — The intervention was developed based on the Behaviour Change Wheel, aiming to increase participants' capability, opportunity, and motivation to engage in physical activity. It consisted of three components: printed materials, group workshops, and an online social media support group.
  * The printed materials included three parts: a culturally appropriate core booklet; the Chinese version of the Otago home exercise booklet, and a physical activity logbook.
  * Participants were invited to attend three workshops over a 12-week period, scheduled every four weeks. The workshops were designed to reinforce the content of the booklets and included presentations, group exercises, and group discussions.
  * Participants were also invited to join a study-specific social media support group via WeChat or WhatsApp, depending on their preference. These groups provided peer support, opportunities to share physical activity goals and progress, and motivational messages and reminders from the researcher.
  Arms: The culturally appropriate physical activity promotion strategies
Behavioral: WHO leaflet group (control) — In the control group, participants received a printed leaflet outlining World Health Organization (WHO) physical activity recommendations for older adults. Participants were encouraged to follow these guidelines, including 150-300 minutes of moderate-intensity or 75-150 minutes of vigorous-intensity aerobic activity per week, along with strength and balance exercises twice weekly, at a time and place convenient to them. No additional support was provided.
  Arms: WHO physical activity guideline group

SUMMARY:
The goal of this study was to explore the feasibility and acceptability of conducting a feasibility randomised controlled trial of culturally appropriate physical activity (PA) promotion strategies among older Chinese adults living in the UK.

The main questions the study aimed to answer were:

Whether older Chinese adults in the UK were willing to take part in the study and to be randomly assigned to a group

Whether participants were willing to remain in the study for its full duration

Whether participants were willing to engage with the PA promotion strategies, including attending workshops, using a logbook, wearing a pedometer, and joining a social media support group

Whether participants found the PA promotion strategies and outcome measures acceptable

Whether physical activity, physical function, and quality of life showed changes in the intervention and control groups

Researchers compared the culturally appropriate PA promotion strategies with a World Health Organization (WHO) PA recommendation leaflet. The study lasted 18 weeks, including a 12-week intervention and a 6-week follow-up.

Participants in the intervention group received culturally appropriate PA promotion materials, including booklets, workshops, a social media support group, a resistance band for strength and balance exercises, and a pedometer.

Participants in the control group received a WHO PA information leaflet and a pedometer.

Participants in both groups completed data collection at three time points. At each time point, participants were asked to wear a pedometer for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or above;
* Self-identified as Chinese ethnicity;
* Speaking either Cantonese, Mandarin and/or English;
* Able to read and write Chinese or English;
* No time requirement for their stay in the UK, but they should have settled in the UK as residents and not as tourists.
* Self-report not meeting the PA guidelines for older adults (engaging in less than 150 minutes of moderate-level PA each week and performing balance, strength, and flexibility exercises less than twice a week);
* Self-report being able to walk around at home independently;
* Can provide informed consent.

Exclusion Criteria:

* Those who self-report that they already meet the PA guidelines (engaging in more than 150 minutes of moderate-level PA each week and performing balance, strength, and flexibility exercises more than twice a week), as this study focuses on older Chinese adults with insufficient PA.
* Those who plan to be away from Manchester for more than 2 months during the intervention period.
* Participants with diseases where exercise is contraindicated will be excluded to ensure the safety of the participants. A self-reported approach will be used to identify these conditions, including cognitive impairment, as it is considered more acceptable by PCIE participants than formal assessments such as the MMSE (Mini-Mental State Examination), which were viewed as burdensome. To mitigate potential bias, the research team will monitor participants throughout the study. Participants who show signs of impairment after giving consent, such as difficulty completing data collection or following instructions, will be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  We aimed to recruit at least 30 participants within eight weeks. Detailed records were kept of the total number of potential participants approached by the researcher, the number of participants who attend the screening, and the number of participants who are ultimately included in the study.
Compliance rate and follow-up rate. | 18 weeks
  Participants were not fully withdrawn from the study solely due to discontinuation of or noncompliance with the intervention. For example, participants could choose to stop attending workshops or participating in the social media group while still remaining willing to complete data collection activities. Alternatively, participation could be discontinued based on clinical judgment. Every effort was made to collect as much data as possible to maintain the integrity of the study. Reasons for participants' exit from the trial were recorded separately.
Adherence | 12 week
  In this study, adherence was mainly assessed by the number of workshops attended by the participants.
Acceptability | 12 to 18 week
  Qualitative interviews. At the end of the study, about 50% of participants (including those who withdraw from the trial) was invited for follow-up interviews.

SECONDARY OUTCOMES:
Subjective measures of physical activity | Baseline, 12-week and 18-week
  Subjective measurement was conducted using the Chinese version of the Physical Activity Scale for the Elderly (PASE).
Objective measures of physical activity | baseline, 12-week and 18-week
  A pedometer (Realalt 3DTriSport 3D Pedometer; 3DTriSport Pedometer for Walking with Clip and Lanyard - Realalt) was used to monitor participants' PA level (i.e., step counts).
COM-B questionnaires | Baseline, 12-week and 18-week
  Brief COM-B questionnaires was used to assess the perceived capability, opportunity and motivation for PA behaviour among older Chinese adults in the UK.
Physical Function | Baseline, 12-week and 18-week
  The Short Physical Performance Battery (SPPB) will be used to assess the potential change of physical function
Health-related quality of life | Baseline, 12-week and 18-week
  The CASP-12 (Control, Autonomy, Self-realisation, and Pleasure-12) questionnaire was used to measure older adults' health-related quality of life
Adverse events | Whole study period-18 weeks
  A safety reporting protocol was followed for managing related and unexpected serious adverse events (SAEs) and directly attributable adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Manchester, Manchester, Great Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request

REFERENCES:
- See also: Published protocol — https://link.springer.com/article/10.1186/s40814-025-01693-7